CLINICAL TRIAL: NCT04059042
Title: Analgesic Effect of Music Listening During Pain Elicitation in Fibromyalgia
Acronym: FMMusic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research activities suspended March 2020 due to COVID-19 pandemic.
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Rebecca Lepping, Ph.D., Senior Scientist, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00144158
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia
Keywords: Pain; Music; Analgesia
MeSH Terms: conditions — Fibromyalgia; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Two-arm (Music, Nature Sounds) parallel randomized controlled pilot study in patients with fibromyalgia with between-subject counterbalanced repeated measure control (Silence). The primary outcome measure will be pain threshold and tolerance as measured by the quantitative sensory testing (QST) battery.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Personnel who interact directly with the study subjects (either human or non-human subjects) will not be aware of the assigned treatments. (Commonly known as "double blind") Personnel who analyze the data collected from the study are not aware of the treatment applied to any given group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): The investigators will manipulate the audio environment the participant experiences 10 minutes before and throughout pain threshold testing (~1 hour). All participants will have one testing session with silence (testing as usual control). On the other testing session, participants will hear music.
  The musical selections will be professional recordings of instrumental Classical music selected by the researcher. All participants will hear the same pieces in the same order. Instrumentation ranges from piano solo to full orchestra, but they are without lyrics or heavy percussion. Pitch ranges across the pieces, but is standard across participants and not controlled by either the participant or the researcher. Tempo for all of the pieces is slow (~60 beats per minute). The pieces are in either major keys or minor keys, but all consist primarily of consonant harmonies and sustained melodic phrases. Participants will control the volume to their individual comfort level.
  Interventions: Behavioral: Music Listening
- Nature Sounds (Placebo Comparator): The investigators will manipulate the audio environment the participant experiences 10 minutes before and throughout pain threshold testing (~1 hour). All participants will have one testing session with silence (testing as usual control). On the other testing session, participants will hear nature sounds.
  Professional recordings of nature sounds selected by the researcher without added music will be used as the active placebo control condition. All participants will hear the same recording. This active control condition will allow for non-musical analgesic effects, such as distraction, to be controlled in the experimental design. Participants will control the volume to their individual comfort level.
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Music Listening — Participants will have pain threshold testing while listening to silence, music, or nature sounds.

SUMMARY:
Patients with fibromyalgia (FM) are more sensitive to things that cause pain. Music lowers self-reported pain in patients with chronic pain. The investigators are able to measure pain sensitivity and pain tolerance using tools that cause pain and give accurate measurements of how much pressure is put on the body (QST). Previous studies have shown that after a few minutes of listening to music patients with FM have less self-reported pain, can get up and move from sitting more quickly, and have more activity in part of the brain that tells the body to stop sending pain signals. The investigators will study 40 patients with FM using the QST tools. All patients will have testing done as usual, with no sound. Then half of the patients will have testing done while listening to instrumental Classical music, and the other half will have testing done while listening to nature sounds. The investigators will test 1) whether listening to anything lessens pain compared to listening to nothing at all; and 2) whether listening to music lessens pain more than listening to nature sounds. Our study will be the first to study whether objectively measured pain sensitivity is less while listening to music in these patients.

DETAILED DESCRIPTION:
Fibromyalgia can be thought of as a centralized pain state where pain is manifested and experienced in different body regions at different times. Individuals with centralized pain feel more pain than would be normally expected based on the level of nociceptive input. Music has previously been shown to have a positive effect on pain, anxiety, and depression in chronic pain patients. However, the impact of music listening on objective measures of pain sensitivity in patients with chronic pain have not yet been described. The goal of this pilot study is to begin to understand the possible analgesic effects of music listening on objective measures of pain sensitivity in patients with fibromyalgia. Previous studies in patients with FM have shown that patients have reduced self-reported pain, increased mobility, and activation of the descending pain modulatory system in the brain after even a short, 5 to10-minute music listening intervention. Our proposed study will be the first to investigate whether objectively measured pain sensitivity is reduced by music listening in these patients.

This two-arm parallel randomized controlled pilot study will enroll 40 patients with fibromyalgia. Patients' pain thresholds and sensitivity will be measured using a battery of quantitative sensory tests (QST). All patients will have two testing sessions: one under testing as usual conditions with no-sound, and one while listening to either instrumental Classical music, selected by the researchers with careful consideration of the musical characteristics, or a nature sound placebo control condition. This careful experimental design will allow us to test whether music listening elicits greater analgesic effects over simple auditory distraction. To minimize potential bias the investigators will employ sound cancelling headphones and randomization of conditions so that the researcher collecting the QST measures will be blinded to whether the patient is hearing music, nature sounds, or nothing. The proposed study is significant as it will identify whether music listening has an analgesic effect during pain threshold and tolerance testing for patients with FM that supercedes any effect of auditory distraction. Results from the proposed study may provide objective evidence that music listening objectively improves analgesia and pain management and thus could be considered therapeutic during situations where acute pain is expected

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and speak English to allow for written informed consent, phenotyping, and patient- reported outcomes measures
* Willingness to refrain from alcohol and nicotine on day of QST
* Willingness to refrain from physical activity or exercise that would cause muscle and/or joint soreness for 48 hours prior to testing (routine exercise or activity that does not lead to soreness is acceptable)
* The investigators will attempt to recruit individuals with no chronic daily use of adjunctive pain medications, including tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors, and gabapentinoids as these drugs can influence QST findings, or have individuals be weaned off of these meds at least two weeks prior to being studied. If the investigators do need to allow individuals into these cohorts while on such medications because of pragmatic issues, this information will be recorded and patients will be asked to remain on a stable dose for at least two weeks prior to QST assessments.

Exclusion Criteria:

* Individuals receiving or applying for compensation or disability and other aspects associated with potential secondary gain
* Inability to provide written informed consent
* Peripheral neuropathy or loss of sensation in the upper or lower extremities which would preclude QST testing
* Severe physical impairment (e.g., blindness, deafness, paraplegia)
* Co-morbid medical conditions that may significantly impair physical functional status (e.g., history of non- skin malignancy, or autoimmune disorder)
* Illicit drug or unreported opioid use (unreported opioid use would be considered opioid abuse and thereby excluded)
* Medical or psychiatric conditions that in the judgment of study personnel would preclude participation in this study (e.g., malignancy, psychosis, suicidal ideation)
* Pregnant or nursing
* Liver failure
* Self-reported liver cirrhosis
* Self-reported hepatitis
* Severe Cardiovascular disease (examples: history of myocardial infarction, unstable angina, severe coronary artery disease, congestive heart failure, or severe valvular abnormalities) that are self-reported by patient or by medical record
* Average daily opioid dosing of >15 mg oral morphine equivalents preoperatively (e.g., > two 5 mg oxycodone tablets/day or > three 5 mg hydrocodone tablets/day). Conversions will be made based on well-accepted conversion tools used previously. The rationale to include some patients taking low dose opioids is to enhance the generalizability of the findings (opioids are common in patients with many pain states), while not causing confounding by including patients on very high doses of opioids which may be a cause of opioid induced hyperalgesia which closely resembles central sensitization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Lepping, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Open Science Framework Registration — http://osf.io/84baz

RESULTS

PARTICIPANT FLOW:
Groups:
- Music: The investigators will manipulate the audio environment the participant experiences 10 minutes before and throughout pain threshold testing (~1 hour). All participants will have one testing session with silence (testing as usual control). On the other testing session, participants will hear music.
  The musical selections will be professional recordings of instrumental Classical music selected by the researcher. All participants will hear the same pieces in the same order. Instrumentation ranges from piano solo to full orchestra, but they are without lyrics or heavy percussion. Pitch ranges across the pieces, but is standard across participants and not controlled by either the participant or the researcher. Tempo for all of the pieces is slow (~60 beats per minute). The pieces are in either major keys or minor keys, but all consist primarily of consonant harmonies and sustained melodic phrases. Participants will control the volume to their individual comfort level.
  Music Listening: Participants will have pain threshold testing while listening to silence, music, or nature sounds.
- Nature Sounds: The investigators will manipulate the audio environment the participant experiences 10 minutes before and throughout pain threshold testing (~1 hour). All participants will have one testing session with silence (testing as usual control). On the other testing session, participants will hear nature sounds.
  Professional recordings of nature sounds selected by the researcher without added music will be used as the active placebo control condition. All participants will hear the same recording. This active control condition will allow for non-musical analgesic effects, such as distraction, to be controlled in the experimental design. Participants will control the volume to their individual comfort level.
  Music Listening: Participants will have pain threshold testing while listening to silence, music, or nature sounds.
Period: Overall Study
Arm/Group | Music | Nature Sounds
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music | Nature Sounds | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.18 (13.86) | 40.28 (9.93) | 44.24 (11.97)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 9
Dominant Hand - Right [Count of Participants; unit: Participants] | 4 | 5 | 9
Education [Count of Participants; unit: Participants]
  High school/GED | 0 | 0 | 0
  Some College | 1 | 1 | 2
  Technical/Associate's degree | 0 | 1 | 1
  Bachelor's degree | 0 | 2 | 2
  Advanced/professional degree | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain Threshold Summation
Description: Pain threshold summation as measured by the quantitative sensory testing (QST) battery. Pain is rated subjectively on a 0-100 scale with 0 being no pain and 100 being the worst pain imaginable. Summation is calculated as the difference in pain score between a single stimulus and a series of 10 stimuli with larger values indicating more severe summation.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a 100 point scale
Arm/Group | Music | Nature Sounds
Number analyzed (Participants) | 4 | 5
units on a 100 point scale
  Audio | 20.25 (14.29) | 4.13 (5.60)
  Silence | 20.17 (13.14) | 9.40 (7.44)
Statistical Analysis 1: Comparison: Music vs Nature Sounds; Test type: Equivalence — Between-session pain measures were assessed with related-samples Wilcoxon signed-rank tests (Audio minus Silence). Data were not normally distributed so nonparametric tests were used; p = .0051, Wilcoxon (Mann-Whitney); Z score = 39.00
Statistical Analysis 2: Comparison: Music vs Nature Sounds; Test type: Equivalence — Between-session change scores were calculated per participant as Audio minus Silence and compared between groups with independent samples Mann-Whitney U-tests. Data were not normally distributed so nonparametric tests were used; p = 0.03, Wilcoxon (Mann-Whitney); Z score = 19.00

2. Primary Outcome: Pain Tolerance
Description: Pain tolerance as measured by the quantitative sensory testing (QST) battery. Pain is rated subjectively on a 0-100 scale with 0 being no pain and 100 being the worst pain imaginable. Tolerance is the pressure (kg/cm2) at which participants rated pain in their non-dominant thumb at 70 out of 100.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Music | Nature Sounds
Number analyzed (Participants) | 4 | 5
kg/cm2
  Audio | 4.12 (1.02) | 5.17 (0.85)
  Silence | 4.18 (1.00) | 5.05 (0.94)
Statistical Analysis 1: Comparison: Music vs Nature Sounds; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.59, Wilcoxon (Mann-Whitney); Z score = 18.00
Statistical Analysis 2: Comparison: Music vs Nature Sounds; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.41, Wilcoxon (Mann-Whitney); Z score = 14.00

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Music | Nature Sounds
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Music (N=5) | Nature Sounds (N=5)
Incidental Finding (Cardiac disorders) | 1 (1) | 0 (0) — Incidental cardiac finding during research ECG

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of participants analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04059042/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT04059042/ICF_001.pdf